CLINICAL TRIAL: NCT04514731
Title: Neuroendocrine Changes Associated With Magnesium Sulfate Administration in Surgical Patients
Brief Title: Magnesium Sulfate and Neuroendocrine Hormone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Jung Shin, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B-2008/631-002
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Arthropathy of Knee; Magnesium Sulfate; Cortisol; Dehydroepiandrosterone
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Experimental): Patients in the magnesium sulfate group received magnesium sulfate 50 mg/kg for 15 minutes after spinal anesthesia and then 15 mg/kg/hour by continuous intravenous infusion until the end of surgery
  Interventions: Drug: Magnesium sulfate
- Group S (Placebo Comparator): Patients in the saline group received the same volume of isotonic saline over the same period with magnesium infusion protocol
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: Magnesium sulfate — Magnesium group receives magnesium sulfate (50 mg/kg) in 100 mL of isotonic saline over 15 minutes after spinal anesthesia, followed by a continuous magnesium sulfate infusion (15 mg/kg/hour) until the end of surgery.
  Arms: Group M
Drug: Isotonic Saline — Isotonic saline group receives the same volume of isotonic saline, administered according to the same methods as in the magnesium group.
  Arms: Group S

SUMMARY:
Total knee arthroplasty is a procedure that relieves pain in patients with severe symptomatic osteoarthritis, but it can be associated with postoperative pain, which hinders recovery. In the previous study, we reported evidence of increased pain in patients undergoing staged total knee arthroplasty, in whom the second operated knee had greater sensitivity (tertiary hyperalgesia) as a result of the surgical injury to the first operated knee.

Magnesium sulfate is an effective analgesic adjuvant for postoperative pain. Its analgesic property seems to be associated with the regulation of calcium influx into the cells, or antagonism of N-methyl-D-aspartate receptors in the central nervous system. Additionally, magnesium is known to have an anti-inflammatory effect. Inflammatory state may accompany with pain via peripheral or central sensitization.

Recently, we reported that magnesium sulfate effectively attenuates not only postoperative pain but also increased pain intensity without serious adverse effects in the bilateral staged total knee arthroplasty. However, the exact mechanism regarding these effects of magnesium sulfate remains unclear.

In the present study, we will investigate the analgesic mechanism of magnesium sulfate via analysis of endocrine neurosteroid levels in patients undergoing bilateral staged total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo staged bilateral total knee arthroplasty
* Spinal anesthesia
* American Society of Anesthesiologists physical status 1 and 2

Exclusion Criteria:

* Patients who undergo unilateral total knee arthroplasty
* General anesthesia
* Musculoskeletal disease
* Hypermagnesemia
* Atrioventricular block
* Previous history of administration of calcium channel blockers

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
The profiles of cortisol in the saliva | From the evening (21:00) before the operation day to the morning (60 minutes after wake-up) of the operation day, for each stage of the operation
  The cortisol concentrations in the saliva, at the evening before the operation (21:00~22:00), just after wake-up in the morning of the operation day, and 30 and 60 minutes after wake-up
The profiles of dehydroepiandrosterone (DHEA) in the saliva | From the evening (21:00) before the operation day to the morning (60 minutes after wake-up) of the operation day, for each stage of the operation
  The DHEA concentrations in the saliva, at the evening before the operation (21:00~22:00), just after wake-up in the morning of the operation day, and 30 and 60 minutes after wake-up

SECONDARY OUTCOMES:
Postoperative pain | Postoperative 24 hour
  Numerical rating scale pain score
Postoperative pain | Postoperative 48 hour
  Numerical rating scale pain score
Patient controlled analgesia (PCA) | Postoperative 24 hour
  Amounts of PCA consumption
Patient controlled analgesia (PCA) | Postoperative 48 hour
  Amounts of PCA consumption
Nausea | Postoperative 24 hour
  Incidence of nausea
Nausea | Postoperative 48 hour
  Incidence of nausea
Vomiting | Postoperative 24 hour
  Incidence of vomiting
Vomiting | Postoperative 48 hour
  Incidence of vomiting
Anti-emetics | Postoperative 24 hour
  Amounts of anti-emetics consumption
Anti-emetics | Postoperative 48 hour
  Amounts of anti-emetics consumption

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Jung Shin, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea